CLINICAL TRIAL: NCT00409045
Title: Evaluation of Obstructive Sleep Apnea as a Risk Factor for Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: Atlantic Health System (Other)
Other Study IDs: R05-08-002; Sleep Apnea
Record Dates: First submitted 2006-12-06; First posted 2006-12-08 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-10

CONDITIONS: Obstructive Sleep Apnea; Pulmonary Embolism
Keywords: Obstructive Sleep Apnea; Pulmonary Embolism; male and female patients suspected of having a pulmonary embolism.
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pulmonary Embolism

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
we evaluate the presence of OSA in patients that have a computed tomography (CT) of the chest to rule out pulmonary embolism (PE) to determine if OSA constitutes an independent risk factor for PE.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients age 18 years and older with suspected PE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male and female patients age 18 years and older
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2005-11; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Epstein, MD, Principal Investigator — Atlantic Health System - Morristown Memorial Hospital
Locations (1):
- Morristown Memorial Hospital, Morristown, New Jersey, United States

REFERENCES:
- [Derived] Epstein MD, Segal LN, Ibrahim SM, Friedman N, Bustami R. Snoring and the risk of obstructive sleep apnea in patients with pulmonary embolism. Sleep. 2010 Aug;33(8):1069-74. doi: 10.1093/sleep/33.8.1069. PMID 20815188